CLINICAL TRIAL: NCT03725189
Title: Pilot Study of the Effect of Physical Activity on Pulse Waveform Monitored by a Novel Photophlethysmographic Device
Brief Title: Photophlethysmography Evaluation of Pulse Waveform
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Taiwan Normal University (Other)
Responsible Party: Principal Investigator, Kakit P. Hui, MD, Principal Investigator, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 00000
Record Dates: First submitted 2018-10-11; First posted 2018-10-30 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Healthy
Keywords: Photophlethysmograph; device; pulse waveform

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PPG Group (Experimental): Testing of PPG device in healthy adult population doing cardiovascular exercise
  Interventions: Device: PPG during exercise

INTERVENTIONS:
Device: PPG during exercise — PPG use for pulse waveform evaluation of healthy exercise group

SUMMARY:
Aim 1. To explore a novel, non-invasive PPG technology for purposes of monitoring heart rate variability and pulse waveform by harmonic resonance analysis.

Aim 2. To analyze collected data to determine whether it provides useful information about other measures of underlying health.

DETAILED DESCRIPTION:
The proposed study will first investigate whether a novel PPG device will be able to measure the harmonic-analysis indexes of the blood pressure waveform (BPWs) to provide information about arterial pulse transmission (by monitoring arterial pulse waveform, Cn) and cardiovascular regulatory activities (by monitoring coefficients of variation, CVn).

Secondarily, data on Cn and CVn could be useful for detecting the arterial elastic properties induced by external stimulation such as exercise, cold stimulation, mental stress, acupuncture, medications such as antihypertensive drugs, or pathological factors such as metabolic syndrome, and breast cancer. The collected data may thus provide information about underlying health.

Photoplethysmography (PPG) is a non-invasive optical technique for evaluating the pulse and hemodynamic changes in frequency. The device obtains a volumetric measurement of an organ via optical illumination (e.g LED). PPG has been used to determine the PaO2, heart rate, and blood pressure (systolic blood pressure, SBP and diastolic blood pressure, DBP) at fingertip and harmonic proportion at fingertip or from the radial artery waveform at the wrist.

However, to the investigator's knowledge, this is the first preliminary study to determine the effects of physical activity on harmonic proportion evaluating by PPG at fingertip. Ultimately, this data may help to develop a non-invasive, external device that could rapidly detect information about cardiovascular and underlying health.

ELIGIBILITY:
4) Inclusion criteria:

1. Ability to understand consent (no proxy consent) in English or Chinese.
2. Self-Reported ability to undertake a 20 minute cycling activity at 60-70% exercise intensity.
3. Ability and willingness to abstain from use of medications for three days preceding cycling activity, smoking/intense exercise/alcohol for 12 hours preceding cycling activity, and caffeine intake for 4 hours preceding cycling.

5) Exclusion criteria:

1. Inability to finish a 20 min cycling activity in 60-70% exercise intensity.
2. Adverse reaction to adhesive tape.
3. Raynaud's phenomenon
4. Angina or recent myocardial infarction (previous 6 months)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Harmonic measures (C1-C10) by PPG device | 70 minutes on Day 1 for resting, exercise, and cool down measurements
  C1-C10 by PPG device

SECONDARY OUTCOMES:
Demographic Information | Day 1
  Collected from patients by questionnaire
General health | Day 1
  General health questionnaire
Weight | Day 1
  Weight
Height | Day 1
  Height
Body mass index (BMI) | Day 1
  Body mass index (BMI)
Diastolic blood pressure (DBP) | 70 minutes on Day 1 for resting, exercise, and cool down measurements
  iHealth Feel Wireless blood pressure monitor
Systolic blood pressure (SBP) | 70 minutes on Day 1 for resting, exercise, and cool down measurements
  iHealth Feel Wireless blood pressure monitor
HRV measures (SDNN, HF, LF and HF/LF parameters) | 70 minutes on Day 1 for resting, exercise, and cool down measurements
  emWave Pro plus, SDNN indicates standard deviation of normal to normal R-R intervals, where R is the peak of a QRS complex (heartbeat). LF and HF represent power in low- and high-frequency ranges
Heart rate and Heart Rate Variation | 70 minutes on Day 1 for resting, exercise, and cool down measurements
  emWave Pro Plus

CONTACTS AND LOCATIONS:
Overall Officials: Ka-Kit Hui, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- National Taiwan Normal University, Taipei, Taiwan